CLINICAL TRIAL: NCT07189936
Title: Mechanism of Isolevuglandin-Protein Adduct Formation in Persistent Immune Activation in Long COVID POTS
Brief Title: Effect of 2-HOBA in Persistent Immune Activation in Long COVID POTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2-HOBA in POTS
Record Dates: First submitted 2025-09-22; First posted 2025-09-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute COVID-19 Syndrome; Postural Tachycardia Syndrome (POTS); SARS CoV 2 Infection; Long COVID19
Keywords: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: A two-parallel arm, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A licensed MTI BioTech (MTI) to develop 2-HOBA. MTI will provide 2-HOBA and matching placebo capsules for the study . Capsules will be shipped to the Vanderbilt Investigational Drug Services (IDS) for use in this trial. The IDS will be responsible for storage, and labeling of 2-HOBA and matching placebo, and for maintaining accurate drug storage and dispensing logs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Levels of circulating monocyte/ T cell doublets, and inflammatory cytokines in 2 HoBA Vs Placebo (Placebo Comparator): to test the effect of 28-day treatment with Iso-LG-adduct scavenger, 2-hydroxybenzylamine (2-HOBA) versus placebo on circulating monocyte/ T cell doublets (CD14+CD3+) , and inflammatory cytokines
  Interventions: Drug: To Measure levels of circulating monocyte/ T cell doublets at Baseline; Drug: To measure levels of circulating monocyte/ T cell doublets after 28 days of 2 HOBA treatment; Drug: To measure levels of circulating monocyte/ T cell doublets after 28 days of Placebo treatment
- Effect of 2HOBA on Splanchnic venous capacitance and compare with placebo group on POTS patients (Placebo Comparator): To test the hypothesis that IsoLG-adducts directly contribute to splanchnic vasodilation, by assessing changes in splanchnic venous capacitance with 2-HOBA treatment at head up Tilt
  Interventions: Diagnostic Test: To Measure Splanchnic venous capacitance after 28 days of Treatment with 2HOBA; Diagnostic Test: To Measure Splanchnic venous capacitance after 28 days of Treatment with Placebo
- Effect of 2HOBA on Orthostatic Tachycardia compare with placebo group during 30 minutes head up tilt (Active Comparator): To test that IsoLG-adducts directly effect Orthostatic tachycardia in LCPOTS, during 30-minute head-up tilt.
  Interventions: Diagnostic Test: To Measure Orthostatic Tachycardia after 28 days of Treatment with 2HOBA; Diagnostic Test: To Measure Orthostatic Tachycardia after 28 days of Treatment with Placebo

INTERVENTIONS:
Drug: To Measure levels of circulating monocyte/ T cell doublets at Baseline — To determine the levels of circulating monocyte/ T cell doublets on all the LCPOTS subjects
  Arms: Levels of circulating monocyte/ T cell doublets, and inflammatory cytokines in 2 HoBA Vs Placebo
Drug: To measure levels of circulating monocyte/ T cell doublets after 28 days of 2 HOBA treatment — Subjects will be randomized 1:1 to 2-HOBA or matching placebo. The levels of circulating monocyte/ T cell doublets (immune burden) after 28 days of 2 HOBA treatment
  Arms: Levels of circulating monocyte/ T cell doublets, and inflammatory cytokines in 2 HoBA Vs Placebo
Drug: To measure levels of circulating monocyte/ T cell doublets after 28 days of Placebo treatment — The levels of circulating monocyte/ T cell doublets (immune burden) after 28 days of 2 HOBA treatment and compare it to the placebo arms
  Arms: Levels of circulating monocyte/ T cell doublets, and inflammatory cytokines in 2 HoBA Vs Placebo
Diagnostic Test: To Measure Splanchnic venous capacitance after 28 days of Treatment with 2HOBA — We will Measure changes in Splanchnic venous capacitance after 28 days of Treatment with 2HOBA and compare it with baseline during 30 Mins head up tilt . All the LCPOTS subjects will be randomized 1:1 to 2-HOBA or matching placebo
  Arms: Effect of 2HOBA on Splanchnic venous capacitance and compare with placebo group on POTS patients
Diagnostic Test: To Measure Splanchnic venous capacitance after 28 days of Treatment with Placebo — We will Measure changes in splanchnic venous capacitance during 30 mins head up tilt ,after 28 days of Treatment with Placebo, we will compare it to the subjects who received 2 HOBA for 28 days
  Arms: Effect of 2HOBA on Splanchnic venous capacitance and compare with placebo group on POTS patients
Diagnostic Test: To Measure Orthostatic Tachycardia after 28 days of Treatment with 2HOBA — To Measure changes in Orthostatic Tachycardia after 28 days of Treatment with 2HOBA at 30 minutes of head up Tilt
  Arms: Effect of 2HOBA on Orthostatic Tachycardia compare with placebo group during 30 minutes head up tilt
Diagnostic Test: To Measure Orthostatic Tachycardia after 28 days of Treatment with Placebo — To Measure changes in Orthostatic Tachycardia after 28 days of Treatment with Placebo at 30 minutes of head up Tilt and compare it with the subjects who received 28 days of 2HOBA
  Arms: Effect of 2HOBA on Orthostatic Tachycardia compare with placebo group during 30 minutes head up tilt

SUMMARY:
Long COVID is defined by a range of symptoms affecting multiple organs that persist for more than three months following an acute SARS-CoV-2 infection. Approximately 7% of individuals who recover from SARS-Cov-2 infection develop Long COVID.

Long COVID Postural Orthostatic Tachycardia Syndrome (LCPOTS) symptoms include fatigue, exercise intolerance, orthostatic intolerance, syncope, and heightened orthostatic tachycardia.

Research has found that decreased parasympathetic activity in LCPOTS increases the production of highly immunogenic neoantigens Isolevuglandins (IsoLG-adducts). IsoLG-adducts induce formation of circulating monocyte/T cell complexes(doublets) leading to the persistent and unresolved immune response that continues after the initial infection.

The purpose of the this research, is to study the effects of 2-hydroxybenzylamine (2-HOBA), an Iso-LG-adduct scavenger, its effects in immune markers and compare it with Placebo

DETAILED DESCRIPTION:
Background:

Decreased parasympathetic activity is present in LCPOTS; this system is an important modulator of NAPDH oxidase activity because the activation of NADPH oxidase in monocytes promotes superoxide (reactive oxygen species -ROS) production.Oxidative stress occurs when ROS are generated in excess of normal antioxidants. Oxidative stress occurs when reactive oxygen species (ROS) are generated in excess of normal antioxidantsOxidative stress occurs when reactive oxygen species (ROS) are generated in excess of normal antioxidants that can cause harm by having adverse effects on T cell function. Targeting downstream damaging effects of ROS is an attractive alternative.

Rationale and Specific Aims

Reduced parasympathetic activity increases the production of highly immunogenic neoantigens, Isolevuglandins (IsoLG-adducts), through heightened activation of NADPH oxidase. Previous findings demonstrated that the cholinergic enhancer galantamine, reduces NADPH oxidase activation and that vagal stimulation reduces IsoLG-adducts in immune cells of LCPOTs patients.

Immune activation in response to viral or likely self-antigen presentation can induce formation of circulating monocyte/T cell complexes(doublets).The presence of these doublets provides powerful insights into the persistent and unresolved immune response that continues after the initial infection. The preliminary data show that: 1) LCPOTS subjects have markedly increased circulating doublets compared to controls; 2) T cells in these doublets produce higher levels of inflammatory cytokines IL-17A and IFN-ɣ than singlet T cells; and 3) inflammatory cytokines positively associate with the severity of orthostatic tachycardia in LCPOTS.

Monocytes in these doublets exhibit high levels of IsoLGs. These results support the hypothesis that LCPOTS represents a condition of unresolved immune activation due to IsoLG-adducts, which we have shown can act as neoantigens.

Study Aims Aim 1: To test the hypothesis that IsoLG-adducts directly contribute to persistent immune activation as measured by elevated monocyte/T cell doublets in LCPOTS.

For this purpose, the effect of 28-day treatment with Iso-LG-adduct scavenger, 2-hydroxybenzylamine (2-HOBA) versus placebo will be tested on circulating monocyte/ T cell doublets, and inflammatory cytokines.

Aim 2: To test the hypothesis that IsoLG-adducts directly contribute to splanchnic vasodilation, orthostatic tachycardia, and symptom burden in LCPOTS.

Aim 2 will be tested using the same experimental design as Aim 1 but will be focused on assessing changes in splanchnic venous capacitance with 2-HOBA treatment.

The proposed study will determine if IsoLG-adducts contribute to persistent immune activation, increased splanchnic venous capacitance, and orthostatic tachycardia in LCPOTS. The goal is to discover new treatment pathways for this disabling disease.

Study population: Total of 50 LCPOTS patients

Study visits: 3 in person study visits and 1 telemedicine

Study Interventions 2-HOBA: 2-hydroxybenzylamine, an IsoLGs potent scavenger.

Safety of 2-HOBA: 2-HOBA was found to be non-cytotoxic and non-mutagenic. It showed a low risk of QT prolongation. Two phase I studies on healthy subjects showed no serious side effects from 2-HOBA at doses ranging from 50 mg to 825 mg. Adverse events (AEs) reported were minor (e.g., headache, sleepiness, abdominal bloating) and were not dose-dependent.

2-HOBA is considered safe for healthy humans.

Dose: A dose of 500 mg three times daily for 28 day to study 2-HOBA for LCPOTS.

Biostatistical Considerations:

Sample size justification and study power (Aim 1). A mean percent of doublets of 5.37 and an SD of 4.28 for the LCPOTS group and a mean percent of doublets of 1.80 and an SD of 1.15 for the control group. The study is to assess for the primary comparison (2-HOBA vs. placebo). A sample size of 16 completed subjects per study arm will have 85% power to detect a 3.57 clinically meaningful difference, i.e., 5.37 versus 1.80 using a Welch t-test. Assuming a drop-out rate of 11%, we need to enroll 18 subjects to have 16 complete subjects per group. Given that subjects will be randomly assigned to two groups. The total enrollment needs to be 36 LCPOTS patients.

Sample size justification and study power (Aim 2). In a previous study, nitroglycerine produces a change from baseline in the Y-intercept of the P-V relationship of 5.7% with a standard deviation (SD) of 1.8 in healthy subjects. A clinically significant difference in the response to 2-HOBA versus placebo is assumed would be at least 35% of that produced with nitroglycerine, with conservatively slightly larger SD of 2.0. The study needs 19 patients per group to be able to reject the null hypothesis that this response difference is zero with a probability (power) of 85%. The Type I error probability associated with this test of this null hypothesis is 0.05. Assuming an attrition rate of 11%, the study needs 25 patients per treatment group. The total enrollment thus needs to be 50 LCPOTS patients.

Statistical Analyses:

The analysis population includes all randomized participants following intention-to-treat analyses.

Aim 1: For the primary comparison between 2-HOBA and placebo, a linear regression model will be used, with doublets (the primary endpoint) at the end of the 28-day treatment as the dependent variable and group indicator, baseline doublets, and other pre-specified baseline variables (age and sex) as covariates.

Aim 2: For the primary comparison between 2-HOBA versus placebo, a linear regression model will be used where splanchnic venous capacitance (SVC, primary endpoint) at the end 28-day treatment is the dependent variable and group indicator and baseline SVC and age and sex as covariates. For both aims, the null hypothesis of no group difference corresponds to the coefficient for the group indicator, which is zero. Appropriate transformation will be used on the outcome variable for the regression models when the normality assumption is violated. Other secondary endpoints will be analyzed similarly to the primary endpoint. The primary and secondary analyses will be conducted without imputing missing data. To protect privacy, subjects will receive a de-identified code. Data will be stored in a password protected, encrypted, and HIPAA compliant REDCap database.

Data and Safety Monitoring Plan:

Data and Safety Monitoring Officer (DSMO) will meet at least twice a year and review data on AEs, data quality, and study recruitment. Reports will be sent to the IRB and FDA at least yearly. Serious AEs will be reported to the FDA following guidelines using the online reporting portal.

ELIGIBILITY:
Inclusion Criteria:

All participants should meet diagnostic criteria for Long COVID and POTS and as outlined below:

Long COVID (LC) is defined by a range of symptoms affecting multiple organs that persist for more than three months following an acute SARS-CoV-2 infection.

POTS: the presence of chronic symptoms lasting more than 3 months, along with orthostatic tachycardia (a HR increase over 30 bpm upon standing or exceeding 120 bpm without orthostatic hypotension) within 10 minutes upon standing or 75-degree head up tilt.

For patients aged 18 and 21, an increase of more than 40 bpm or a standing HR over 130 bpm will be required for inclusion in the study.

2 Patients need confirmation of POTS diagnosis based on orthostatic vital signs obtained prior to enrollment in the study.

SARS-CoV-2 infection 3 or more months prior identified by the follow signs:

A. Meets the clinical OR epidemiological criteria.

1. Clinical criteria: Acute onset of fever AND cough (influenza-like illness) OR Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general, weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, nausea, diarrhea, anorexia.
2. Epidemiological criteria: Contact of a probable or confirmed case or linked to a COVID-19 cluster; or B. Presents with acute respiratory infection with history of fever or measured fever of ≥ 38°C; and cough; with onset within the last 10 days; and who requires hospitalization); or C. Presents with no clinical signs or symptoms, NOR meeting epidemiologic criteria with a positive professional use or self-test SARS-CoV-2 antigen-Rapid Diagnostic Test.

D. A person with a positive nucleic acid amplification test, regardless of clinical criteria OR epidemiological criteria; or E. Meeting clinical criteria AND/OR epidemiological criteria (See A). With a positive professional use or self-test, SARS-CoV-2 Antigen-Rapid Diagnostic Test.

F. Documented by health care provider in clinical note or encounter.

Exclusion Criteria:

1. Known active acute SARS-Cov-2 infection (4 weeks from onset)
2. Moderate or severe immunocompromised patients,
3. Known history of cardiovascular disease (atrioventricular block (AV block), myocardial infarction, angina, heart failure, pacemaker, stroke, transient ischemic attack within 6 months before enrollment),
4. Uncontrolled hypertension (BP>140/90 despite appropriate treatment);
5. Type 1 or type 2 diabetes mellitus;
6. Impaired hepatic function (AST or ALT greater than 1.5x the upper limit of normal or with total bilirubin ≥1.5mg/dl),
7. Impaired renal function test (eGFR<60 mL/min/1.73m2),
8. Anemia (hemoglobin <10 g/dl),
9. Pregnant or breastfeeding women,
10. Known history of autoimmune disease, steroid use or other immunotherapies,
11. Inability to provide informed consent.

We will also exclude individuals with known allergy sensitivity to components of the study medication, known contraindication to the study interventions, use of central acetylcholinesterase inhibitors (e.g., pyridostigmine, donezepil), aspirin allergy because salicylic acid is a metabolite of 2-HOBA; use of monoamine oxidase inhibitors (MAO-I) because of some inhibition of MAO-A is present in the anticipated therapeutic range of 2-HOBA.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect IsoLG-adducts (2-HOBA) measured by levels of monocyte/T cell doublets in LCPOTS. | Baseline (Day 0) to after 28 days of treatment
  The effect of 28-day treatment with Iso-LG-adduct scavenger, 2-hydroxybenzylamine (2-HOBA) versus placebo on circulating monocyte/ T cell doublets, and inflammatory cytokines and compare it to the placebo
Changes in Splanchnic venous capacitance before and after 28 days of treatment | Day 0- Day 28 days
  Changes in Splanchnic venous capacitance at 30 mins Head up tilt, before and after 28 days of treatment and compare it with 2-HOBA group with placebo group

SECONDARY OUTCOMES:
Measure the effects of 2- HOBA on Orthostatic Tachycardia at HUT | Baseline (Day0) to after 28 days of study medication
  To see the effects of IsoLG-adducts (2-HOBA) on Orthostatic Tachycardia in LCPOTS subjects at 30 mins Head up Tilt (HUT) and compare it with Placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, M.D, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Cyndya Shibao, Nashville, Tennessee, United States